CLINICAL TRIAL: NCT00631696
Title: Prospective Randomized Double-Blind Study Of Sperm Production In Healthy Volunteers Receiving Pregabalin Or Placebo
Brief Title: Evaluation Of Sperm Production With Healthy Male Volunteers Receiving Lyrica Or Placebo
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: A0081104
Record Dates: First submitted 2008-02-15; First posted 2008-03-10 (Estimated); Results first posted 2012-10-24 (Estimated); Last update posted 2021-01-26 (Actual); Status verified 2012-09

CONDITIONS: Healthy
Keywords: Healthy males Human volunteers pregabalin or placebo sperm quality and quantity
MeSH Terms: interventions — Pregabalin

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Pregabalin
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pregabalin — pregabalin 600 mg given twice a day
  Arms: 1
Drug: Placebo — Placebo
  Arms: 2

SUMMARY:
This study is being performed as a Phase IV FDA commitment study and is being powered adequately to assess changes in sperm concentration, FSH and testosterone in healthy male subjects treated with pregabalin as compared to placebo, in addition to confirming lack of effects on sperm motility.

DETAILED DESCRIPTION:
This is a Phase 4 FDA commitment study. The purpose of the study is to evaluate the effects of pregabalin as compared to placebo on sperm concentration in healthy male subjects

ELIGIBILITY:
Inclusion Criteria:

* Healthy 18 to 55 years old males

Exclusion Criteria:

* Screening sperm count <20 x 106/mL; screening sperm motility <50% motile (a+b) or <25% Class "a" motile or screening sperm morphology <30% normal or semen volume <1.5 mL or white blood cell count >1 x 106 /mL on any screening visit sample

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 222 (Actual)
Dates: Start 2008-02; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (12):
- United States (12):
  - Pfizer Investigational Site, Mobile, Alabama
  - Pfizer Investigational Site, Phoenix, Arizona
  - Pfizer Investigational Site, Tarzana, California
  - Pfizer Investigational Site, Ocala, Florida
  - Pfizer Investigational Site, Madisonville, Kentucky
  - Pfizer Investigational Site, Shreveport, Louisiana
  - Pfizer Investigational Site, Ann Arbor, Michigan
  - Pfizer Investigational Site, Minneapolis, Minnesota
  - Pfizer Investigational Site, Las Vegas, Nevada
  - Pfizer Investigational Site, Durham, North Carolina
  - Pfizer Investigational Site, Cumberland, Rhode Island
  - Pfizer Investigational Site, San Antonio, Texas

REFERENCES:
- [Derived] Sikka SC, Chen C, Almas M, Dula E, Knapp LE, Hellstrom WJ. Pregabalin does not affect sperm production in healthy volunteers: a randomized, double-blind, placebo-controlled, noninferiority study. Pain Pract. 2015 Feb;15(2):150-8. doi: 10.1111/papr.12171. Epub 2014 Jan 23. PMID 24450301
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A0081104&StudyName=Evaluation%20Of%20Sperm%20Production%20With%20Healthy%20Male%20Volunteers%20Receiving%20Lyrica%20Or%20Placebo

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study was conducted at 12 centers in the United States between February 2008 and February 2012; 903 participants were screened and 222 were assigned to study treatment.
Groups:
- Pregabalin: Pregabalin 50 milligrams (mg) by mouth (PO) twice a day (BID) starting dose with a 2-week titration followed by a fixed dose of 300 mg PO BID for 10 weeks, a 1 week taper at Week 12, and a 13 week washout period up to Week 26.
- Placebo: Placebo matching pregabalin treatment.
Period: Overall Study
Arm/Group | Pregabalin | Placebo
Started | 112 | 110
Received Study Treatment (Tx) | 111 | 109
Ongoing at Database Release 18Oct2011 | 2 (Completed Tx at time of database release 18Oct2011; included in all analyses.) | 0
Completed | 75 (Completed study at time of database release 18Oct2011.) | 70 (Completed study at time of database release 18Oct2011.)
Not Completed | 37 | 40
Not completed — Entered, not randomized to treatment | 1 | 1
Not completed — Discontinued after database release date | 1 | 0
Not completed — Follow up after database release date | 1 | 0
Not completed — Lost to Follow-up | 7 | 10
Not completed — Withdrawal by Subject | 2 | 9
Not completed — Other | 8 | 8
Not completed — Protocol Violation | 9 | 9
Not completed — Study terminated by sponsor | 3 | 3
Not completed — Adverse Event | 5 | 0

BASELINE CHARACTERISTICS:
Groups:
- Pregabalin: Pregabalin 50 mg PO BID starting dose with a 2-week titration followed by a fixed dose of 300 mg PO BID for 10 weeks, a 1 week taper at Week 12, and a 13 week washout period up to Week 26.
- Total: Total of all reporting groups
Arm/Group | Pregabalin | Placebo | Total
Number analyzed (Participants) | 111 | 109 | 220
Age, Customized [Number; unit: participants]
  Between 18 and 44 years | 100 | 93 | 193
  Between 45 and 64 years | 11 | 16 | 27
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 111 | 109 | 220

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With a 50 Percent (%) or More Reduction in Sperm Concentration From Baseline (Bsl) to End of Study (EOS)
Description: Baseline is the average of sperm concentrations from semen samples collected on or before Study Day 1. End of study is average of sperm concentrations from semen samples collected at end of washout period (Week 26) following 12 weeks of double-blind treatment. Mean sperm concentration (MSC) of a visit is average of the 2 sperm concentration samples collected at that visit. If sperm concentration was not assessed at Week 26, then the last assessment on or after Week 12 (end of treatment) was used instead. Confidence intervals (CI) based on exact distribution.
Time Frame: Baseline, End of Study (last observation at Week 26 or last assessment on or after Week 12 if no data at Week 26)
Population: Per protocol analysis set: all randomized participants who had ≥8 weeks of study treatment, sperm concentration measurements at or after week 12 window, did not discontinue for site violations, and did not have any major protocol violations. N=number of participants with analyzable data at observation; Last observation carried forward (LOCF).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 65 | 62
percentage of participants | 9.2 [3.46 to 19.02] | 3.2 [0.39 to 11.17]
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Study powered to show non-inferiority (NI) of pregabalin (PGB) to placebo (PBO) on the percentage of participants (N) with a ≥50% reduction in MSC from Bsl to end of washout (Week (Wk) 26, or last assessment on or after Wk 12 if Wk 26 not done). NI to be declared if upper bound of 95% CI for difference between PGB and PBO not >20%. Assuming proportion of N with 50% reduction to be 6% for both groups, sample size N=65 per group would provide >90% power to show NI of PGB to PBO; Test type: Non-Inferiority or Equivalence — A non-inferiority margin of 20% was used to test the hypothesis. The null hypothesis is that the difference (PGB - PBO) in the proportion of participants with ≥50% reduction in sperm concentration is ≥20% and the alternative hypothesis is that the difference in proportion of participant with ≥50% reduction in sperm concentration is <20%; Confidence Interval Approach; percentage difference = 6.0, 95% CI 2-sided [-2.29 to 14.30] — The confidence interval was based on asymptotic normal distribution

2. Secondary Outcome: Change From Baseline in Follicle Stimulating Hormone (FSH) to End of Study (EOS)
Description: FSH minimum normal range 1.4 International units per liter (IU/L) to maximum normal range 18.1 IU/L. End of study was the end of the washout period (Week 26) following 12 weeks of double-blind treatment. If the semen parameter was not assessed at Week 26, then the last assessment on or after Week 12 (end of treatment) was used instead.
Time Frame: Baseline, End of Study (last observation at Week 26 or last assessment on or after Week 12 if no data at Week 26)
Population: Modified intent-to-treat (MITT) population included all randomized participants who received at least 1 dose of study medication (either pregabalin or placebo) and were not discontinued for major violation at the site level. N=number of participants with analyzable data at observation; LOCF.
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 79 | 72
IU/L
  Baseline | 3.17 (1.624) | 3.68 (1.997)
  Change to EOS | 0.14 (0.746) | 0.22 (0.953)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Test type: Superiority or Other; p = 0.3462, ANCOVA — p-value from analysis of covariance (ANCOVA) with treatment and center as main effects and baseline value as covariate in the model; LS Mean Difference = -0.12, 95% CI 2-sided [-0.385 to 0.136] — Least Squares Mean (LS Mean) and 95% CI from ANCOVA with treatment and center as main effects and baseline value as covariate in the model. LS Mean Difference calculated as (Pregabalin - Placebo)

3. Secondary Outcome: Change From Baseline in Follicle Stimulating Hormone (FSH) to Week 26
Description: FSH minimum normal range 1.4 IU/L to maximum normal range 18.1 IU/L. Week 26 was the non-missing value within 134 to 252 days from Study Day 1. If there were multiple observations between the stated study days (all non-missing or a combination of missing and non-missing), then the latest non-missing value was selected for analysis. If all the values within the stated window were missing, then the records were not to be used for Week 26 analysis.
Time Frame: Baseline, Week 26 (last observation in the Week 26 window)
Population: MITT population; N=number of participants (observed cases) with analyzable data at observation.
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 69 | 60
IU/L
  Baseline | 3.20 (1.685) | 3.69 (2.050)
  Change to Week 26 | 0.16 (0.757) | 0.21 (0.949)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Test type: Superiority or Other; p = 0.3652, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.13, 95% CI 2-sided [-0.420 to 0.156] — [estimate comment as in outcome 2, analysis 1]

4. Secondary Outcome: Change From Baseline in Follicle Stimulating Hormone (FSH) to Week 12
Description: FSH minimum normal range 1.4 IU/L to maximum normal range 18.1 IU/L. Week 12 was the last non-missing value within 2 to 133 days from Study Day 1. If there were multiple observations between the stated study days (all non-missing or a combination of missing and non-missing), then the latest non-missing value was selected for analysis. If all the values within the stated window were missing, then the records were not to be used for Week 12 analysis.
Time Frame: Baseline, Week 12 (last observation in the Week 12 window)
Population: MITT; N=number of participants with analyzable data at observation.
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 79 | 72
IU/L
  Baseline | 3.17 (1.624) | 3.68 (1.997)
  Change to Week 12 | -0.05 (0.785) | 0.08 (0.974)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Test type: Superiority or Other; p = 0.1204, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.20, 95% CI 2-sided [-0.464 to 0.054] — [estimate comment as in outcome 2, analysis 1]

5. Secondary Outcome: Change From Baseline in Testosterone to End of Study (EOS)
Description: End of study was the end of the washout period (Week 26) following 12 weeks of double-blind treatment. If the semen parameter was not assessed at Week 26, then the last assessment on or after Week 12 (end of treatment) was used instead.
Time Frame: Baseline, End of Study (last observation at Week 26 or last assessment on or after Week 12 if no data at Week 26)
Population: MITT; N=number of participants with analyzable data at observation; LOCF.
Measure: Mean (Standard Deviation); unit: nanograms per deciliter (ng/dL)
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 79 | 72
nanograms per deciliter (ng/dL)
  Baseline | 518.2 (179.13) | 481.8 (171.07)
  Change to EOS | 10.4 (170.78) | 0.8 (150.64)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Test type: Superiority or Other; p = 0.2875, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = 24.65, 95% CI 2-sided [-20.999 to 70.302] — [estimate comment as in outcome 2, analysis 1]

6. Secondary Outcome: Change From Baseline in Testosterone to Week 26
Description: Week 26 was the non-missing value within 134 to 252 days from Study Day 1. If there were multiple observations between the stated study days (all non-missing or a combination of missing and non-missing), then the latest non-missing value was selected for analysis. If all the values within the stated window were missing, then the records were not to be used for Week 26 analysis.
Time Frame: Baseline, Week 26 (last observation in the Week 26 window)
Population: MITT; N=number of participants with analyzable data at observation.
Measure: Mean (Standard Deviation); unit: ng/dL
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 69 | 60
ng/dL
  Baseline | 517.9 (182.34) | 474.6 (167.09)
  Change to Week 26 | 13.8 (171.37) | 2.6 (146.80)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Test type: Superiority or Other; p = 0.1699, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = 32.93, 95% CI 2-sided [-14.292 to 80.158] — [estimate comment as in outcome 2, analysis 1]

7. Secondary Outcome: Change From Baseline in Testosterone to Week 12
Description: Week 12 was the last non-missing value within 2 to 133 days from Study Day 1. If there were multiple observations between the stated study days (all non-missing or a combination of missing and non-missing), then the latest non-missing value was selected for analysis. If all the values within the stated window were missing, then the records were not to be used for Week 12 analysis.
Time Frame: Baseline, Week 12 (last observation in the Week 12 window)
Population: MITT; N=number of participants with analyzable data at observation.
Measure: Mean (Standard Deviation); unit: ng/dL
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 79 | 72
ng/dL
  Baseline | 518.2 (179.13) | 481.8 (171.07)
  Change to Week 12 | -14.8 (169.56) | 0.0 (123.61)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Test type: Superiority or Other; p = 0.7958, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -6.12, 95% CI 2-sided [-52.804 to 40.558] — [estimate comment as in outcome 2, analysis 1]

8. Secondary Outcome: Change From Baseline in Sperm Motility to End of Study (EOS)
Description: Mean sperm motility (percent motility representing grade a+b [a=sperm with progressive, straight-line motility; b=non-linear motility]) was average of 2 samples collected at that visit. Normal value is ≥50% motility measured within 60 minutes of collection; higher values=greater percentage of sperm with motility. End of study was the end of the washout period (Week 26) following 12 weeks of double-blind treatment. If the semen parameter was not assessed at Week 26, then the last assessment on or after Week 12 (end of treatment) was used instead.
Time Frame: Baseline, End of Study (last observation at Week 26 or last assessment on or after Week 12 if no data at Week 26)
Population: MITT; N=number of participants with analyzable data at observation; LOCF.
Measure: Mean (Standard Deviation); unit: percent motility
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 79 | 73
percent motility
  Baseline | 61.9 (9.98) | 61.4 (8.32)
  Change to EOS | -3.2 (10.57) | -1.8 (7.49)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Test type: Superiority or Other; p = 0.4094, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -1.08, 95% CI 2-sided [-3.645 to 1.494] — [estimate comment as in outcome 2, analysis 1]

9. Secondary Outcome: Change From Baseline in Sperm Motility to Week 26
Description: Mean sperm motility (percent motility representing grade a+b) was the average of 2 samples collected at that visit. Normal value is ≥50% motility measured within 60 minutes of collection; higher values=greater percentage of sperm with motility. Week 26 was average of the last 2 values within window of 134 to 252 days from Study Day 1 and at least 1 of the 2 values was non-missing. If only 1 assessment date within the stated window, Week 26 was the value of that single assessment. If all values within window were missing, the records were not to be used for Week 26 analysis.
Time Frame: Baseline, Week 26 (last observation in the Week 26 window)
Population: MITT; N=number of participants with analyzable data at observation.
Measure: Mean (Standard Deviation); unit: percent motility
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 69 | 60
percent motility
  Baseline | 61.8 (10.46) | 61.2 (8.71)
  Change to Week 26 | -2.6 (9.71) | -1.8 (6.52)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Test type: Superiority or Other; p = 0.9064, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.15, 95% CI 2-sided [-2.649 to 2.352] — [estimate comment as in outcome 2, analysis 1]

10. Secondary Outcome: Change From Baseline in Sperm Motility to Week 12
Description: Mean sperm motility (percent motility representing grade a+b) was average of 2 samples collected at that visit. Normal value is ≥50% motility measured within 60 minutes of collection; higher values=greater percentage of sperm with motility. Week 12 was average of last 2 values within window of 2 to 133 days from Study Day 1 and at least 1 of the 2 values was non-missing. If there was only 1 assessment date within the stated window, then Week 12 was the value of that single assessment. If all the values within the window were missing, then the records were not to be used for Week 12 analysis.
Time Frame: Baseline, Week 12 (last observation in the Week 12 window)
Population: MITT; N=number of participants with analyzable data at observation.
Measure: Mean (Standard Deviation); unit: percent motility
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 79 | 73
percent motility
  Baseline | 61.95 (9.976) | 61.38 (8.316)
  Change to Week 12 | -3.94 (8.570) | -2.71 (8.186)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Test type: Superiority or Other; p = 0.4666, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.86, 95% CI 2-sided [-3.207 to 1.477] — [estimate comment as in outcome 2, analysis 1]

ADVERSE EVENTS:
Time Frame: Treatment emergent Adverse Events are collected from the time of first dose of study treatment through last subject last visit (06 February 2012).
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Pregabalin | Placebo
Serious Adverse Events (participants affected / at risk) | 0/111 | 0/109
Other Adverse Events (participants affected / at risk) | 43/111 | 18/109
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pregabalin (N=111) | Placebo (N=109)
Nausea (Gastrointestinal disorders) | 2 | 4
Fatigue (General disorders) | 5 | 1
Muscle strain (Injury, poisoning and procedural complications) | 4 | 1
Dizziness (Nervous system disorders) | 21 | 1
Headache (Nervous system disorders) | 4 | 5
Paraesthesia (Nervous system disorders) | 4 | 1
Somnolence (Nervous system disorders) | 11 | 5
Euphoric mood (Psychiatric disorders) | 6 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.